CLINICAL TRIAL: NCT00701714
Title: Randomized, Controlled, Double-blind Multicenter Safety Study to Evaluate the Safety and Immunogenicity of Subcutaneous EPO HEXAL vs. ERYPO® in the Treatment of Anemia Associated With Chronic Renal Insufficiency in Predialysis Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: investigation of adverse events
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-22-INJ-17
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Anemia; Chronic Renal Insufficiency
Keywords: Treatment; associated; with CRI
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HX575, EPO HEXAL
  Interventions: Drug: HX575 recombinant human erythropoietin alfa
- 2 (Active Comparator): ERYPO
  Interventions: Drug: ERYPO

INTERVENTIONS:
Drug: HX575 recombinant human erythropoietin alfa — Solution for injection (s.c.)
  Arms: 1
Drug: ERYPO — Solution for injection (s.c.)
  Arms: 2

SUMMARY:
This is a randomized, controlled, double-blind, multicenter multinational safety study involving about 300 predialysis patients aged 18 years or above suffering from anemia.

Symptomatic anemia will be corrected by s.c. application of EPO HEXAL or ERYPO® in order to achieve a hemoglobin target range of 10.0 -12.0 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Known chronic renal insufficiency of at least 4 weeks duration; CKD stage at least 3 or higher
* Male and female patients, age: >=18
* Patients who are naïve to ESA treatment or previously ESA treated after 3 months of ESA-free period (i.v. or s.c.)
* Patients with symptomatic anemia, defined as Hb level below 11.0 g/dL and not lower than or equal to 7.5 g/dL on at least 2 visits during the screening period
* Adequate iron status, serum ferritin >= 100 µg/L or transferrin saturation >= 20%
* Ability to follow study instructions and likely to complete all required visits and compliant with subcutaneous administration
* Written informed consent of the patient.

Exclusion Criteria:

* Anemia of non-renal causes
* Therapy with immunosuppressants (other than corticosteroids for chronic treatment) within 3 months before screening and during the study for patients with renal allograft in place or other chronic conditions (e.g. lupus erythematosus, rheumatic arthritis)
* Patients previously treated with chronic dialysis within the last 6 months (exception: one session of acute dialysis)
* Patients with acute deterioration of renal function during the screening phase according to the investigator's judgment
* Patients receiving any RBC/whole blood transfusion during the screening period
* Primary hematological disorder (e.g. myeloma, myelodysplastic syndrome, sickle cell anemia, hematological malignancy, hemolytic anemia)
* Evidence of uncontrolled diabetes mellitus (HbA1c > 10 % at visit -2)
* Evidence of severe hepatic dysfunction (e.g. ALT and/or AST above 2x upper limit of normal range; or gamma-GT above 3x upper limit of normal range)
* Clinical evidence of current uncontrolled or symptomatic hyperparathyroidism, defined as parathyroid hormone > 500 ng/L at visit -2.
* Uncontrolled hypertension, defined as a systolic blood pressure of >= 160 mmHg and a diastolic blood pressure measurement >= 100 mmHg (average of two values with at least one day between measurements)
* Congestive heart failure and/or angina pectoris [New York Heart Association (NYHA) class III and IV]
* History of stroke or myocardial infarction during the last 6 months prior to visit -2
* Ongoing treatment with phenprocoumon or other cumarin derivates
* Thrombocytopenia (platelet count <100.000/µL) or leucopenia (white blood cell count < 2.000/µL)
* Gastrointestinal bleeding within the last 6 months prior to visit -2 or hemolysis
* Evidence of acute or chronic infection by a C-reactive protein value of > 30 mg/L
* Suspicion or known PRCA (pure red cell aplasia)
* Previously diagnosed HIV or acute hepatitis infection
* History of epilepsy or epileptic seizures or treatment for epilepsy within the past 6 months prior to screening
* Planned major surgery (with expected high blood loss) during the next 3 months or major surgery within the previous 3 months (except laser photocoagulation, access surgery)
* Clinical evidence of active malignant diseases within the last 5 years (except non-melanoma skin cancer)
* Pregnancy, breastfeeding women or women not using a highly effective birth control method (e.g. implants, injectables, combined oral contraceptives, IUD, sexual abstinence, vasectomised partner)
* Known history of severe drug related allergies (e.g. anaphylactic shock)
* Known allergy to one of the ingredients of the test product or hypersensitivity to mammalian-derived products
* Known or suspicion of any non-compliance with respect to subcutaneous treatment
* Simultaneous participation in another clinical study or participation in a study in the month preceding visit-2 or previously randomized in this study
* Participation in another ESA study in the 3 months preceding visit -2
* Any other condition which at the investigator's discretion may put the patient at risk or which may confound the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vetter, Dr., Study Chair — Hexal AG
Locations (123):
- Austria (5):
  - Diakonissen KH Salzburg, Salzburg
  - LKH Steyr, Steyr
  - Krankenanstalt der Stadt Wien, Vienna
  - AKH Wien, Vienna
  - Sozialmedizinisches Zentrum Ost Donauspital, Vienna
- Bulgaria (4):
  - MHAT Pazardijk, Pazardzhik
  - MHAT Sveti Ivan Rilski, Sofia
  - MHAT Stara Zagora, Stara Zagora
  - MHAT "Sv. Anna", Varna
- Czechia (10):
  - Ambulance vnitrního lékarstvi, Brno
  - Nemocnice Kladno, Kladno
  - Litomyslska nemocnice, a.s., Litomyšl
  - Nemocnice s poliklinikou v Novem Jicine, Novi Jicin
  - IKEM, Prague
  - FN Motol, Prague
  - Dialcorp, s.r.o., Praha 4 - Michle
  - Nemocnice Prostìjov, Prostìjov
  - Nemocnice Šternberk, Sternberk
  - Nefrologická a interní amb., Žïár N. Sázavou
- France (2):
  - CHU d'Amiens - Hopital Sud, Amiens
  - CHU de Rouen - Hopital de Bois Guillaume, Bois-Guillaume
- Germany (46):
  - Gesundheitszentrum Alzey, Alzey
  - Studienzentrum Hämatologie / Onkologie / Diabetes, Aschaffenburg
  - Gemeinschaftspraxis Dr. med. Gert-Peter Dragoun, Dr. med Günther Hevendehl, Aschaffenburg
  - Nephrologische Praxis Bad Münder, Bad Münder am Deister
  - Praxis Dr. Scharla, Bad Reichenhall
  - Nephrologisches Zentrum an Stadtkrankenhaus, Bad Wildungen
  - Dialyse-Centrum, Bad Windsheim
  - KfH Kuratorium f. Dialyse und Nierentransplantation e.V., Bergisch Gladbach
  - Schwerpunktpraxis für Diabetologie und Nephrologie, Bernkastel-Kues
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Bischofswerda
  - Dialysepraxis drs. Riedasch/Schreiber, Coesfeld
  - Praxis Dr. Kraatz, Demmin
  - Gemeinschaftspraxis Dr. Steffen & Dr. Perino, Dinkelsbühl
  - Diabetes- und Dialysezentrum Merker, Vogt, Dormagen
  - Gemeinschaftspraxis Karlstraße, Düsseldorf
  - Dialysepraxis Häger, Schanze, Brause, Düsseldorf
  - KfH Kuratorium f. Dialyse und Nierentransplantation e.V., Eberswalde
  - Gemeinschaftspraxis Dr. Spitthöver, Dr. Knee, Dr. Gröschel, Essen
  - Praxis Dr. Zimmermann, Essen
  - Praxis Dr. Lüdemann, Falkensee
  - Dialysepraxis, Friedrichroda
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Fürstenzell
  - Dialysepraxis Barmbek, Hamburg
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Haßfurt
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Heringen
  - Dialysezentrum, Homberg (Efze)
  - Gemeinschaftspraxis und Dialyse, Hürth
  - Dialyseplaxis DR. Rieck, DR. Göbel, DR. Wagner, Krefeld
  - Leipziger Institut für Präventivmedizin, Leipzig
  - Med Center Leipzig, Leipzig
  - GDG Gemeinnützige Dialyse Gesellschaft, Leverkusen
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Ludwigshafen
  - Gemeinschaftspraxis Dres. Leistikow, Hafezi und Sandner, Mannheim
  - Praxis Dr. Schütterle, Marburg
  - Praxis Dr. Vogel-Wagner, Mittweida
  - Praxis Dr. Rose, Pohlmeier und Dr. Lammers, Münster
  - Dialyse Nettetal, Nettetal
  - KfH Kuratorium für dialyse und Nierentransplantation e.V., Nördlingen
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Passau
  - Praxis Dipl. med. Kosch, Pirna
  - Dialysepraxis Dipl. med. Gierak & Dipl. med. Rettig, Quedlinburg
  - Klinik für Nephrologie und Allgemeine Innere Medizin, Solingen
  - Gemeinschaftspraxis Dr. Kirchner und Dr. Menge, Sömmerda
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Straubing
  - Praxis Dr. med. Mauersberger, Villingen-Schwenningen
  - Nephrologische Gemeinschaftspraxis Dr. Rensinghoff & Dr. Becker, Wattenscheid
- India (7):
  - Kamineni Hospitals Ltd., Hyderabaad
  - NIZAM Institute of Medical Sciences, Hyderabaad
  - Bombay Hospital, Indore
  - Monilek Hospital and Research Center, Jaipur
  - Vinaya Hospital & Research Centre, Mangalore
  - Pulse Diagnostix Cardiac and Medical Center, Pune
  - Kerala Institute of Medical Sciences, Trivandrum
- Poland (8):
  - SP ZOZ Miejski Szpital Zespolony, Częstochowa
  - Szpital Wojewódzki w Poznaniu, Poznan
  - Specjalistyczne Centrum Diagnostyczno-Lecznicze Bamberski Dwor (Solumed SC), Poznan
  - Specjalistyczna Przychodnia Lekarska Medikard, Płock
  - NZOZ NEFROLUX Sp. J. Lucjan Sobieraj, Wojciech Kaminski, Siemianowice Śląskie
  - Wojewodzki Szpital Specjalistyczny nr. 1 im. Jozefa Gasinskiego, Tychy
  - Szpital Praski p.w. Przemienienia Panskiego II Oddzia Chorob Wewnetrznych, Warsaw
  - NZOZ Centrum Badan Klinicznych, Wroclaw
- Romania (13):
  - Centrul Medical de Diagnostic si Tratament Ambulator si Medicina Preventiva Bucuresti, Bucharest
  - Institutul National de DiabetNutritie si Boli Metabolice Paulescu, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Universitar Bucuresti, Bucharest
  - Spitalul Clinic Judetean Cluj, Cluj-Napoca
  - County Hospital Deva, Deva
  - Spitalul Clinic CI Parhon Iasi, Iași
  - Dr. Gavril Curteanu Clinical Hospital, Oradea
  - County Hospital Tg Mures, Tg Mures
  - SC Medicali's SRL, Timișoara
  - Emergency Clinical County Hospital, Timișoara
  - Spitalul Judetean Timisoara, Timișoara
  - Policlinica Dr. Citu, Timișoara
- Russia (25):
  - Municipal medical Institution "City Hospital #1", Barnaul
  - State Healthcare Institution "Kemerova Regional Clinical Hospital", Kemerovo
  - Federal State Institution "National Medical Surgery center named after NI Pirogov of Federal Agency of Health Care and Social Development", Moscow
  - State Educational Institution of Higher Professional Education "Moscow State University of Medicine and dentistry of Federal Agency of health Care and Social Development", City Clinical Hospital #23, Moscow
  - Russian University of Peoples Frienship (clinical base: City clinical hospital #53), Moscow
  - State Health Care Institution City Clinical Hospital named after SP Botkin, Moscow
  - State healthcare Institution "Nizhegorodsky Regional Clinical Hospital named after NA Semashko", Nizhny Novgorod
  - State Healthcare Institution "Reoublic Hospital named after VA Baranov", Petrozavodsk
  - Municipal healthcare Institution "City Clinical Hospital #2", Pyatigorsk
  - State Healthcare Institution "Ryazan Regional Cardiological Dispensary", Ryazan
  - State Educational Institution of Higher Professional Education "St. Petersburg State Medical Academy for Postgraduate studies of Roszdrav", Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Mariinsky Hospital", Saint Petersburg
  - State Institution "St. petersburg Clinical research Institute of Emergency Medical Care named after I.I. Dzhanelidze", Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Outpatient Clinic #17", Saint Petersburg
  - State Educational Institution of Higher Professional Education "St. Petersburg State Medical Academy named after I.I. Mechnikov of Roszdrav", Saint Petersburg
  - State Institute St. Petersburg, Saint Petersburg
  - State Educational Institution of Higher Professional Education "St. Petersburg State Medical Institute named after IP Pavlov of Roszdrav", Saint Petersburg
  - State Educational Institution of High Professional Education Saratov State Medical University of Roszdrav, Saratov
  - State Educational Institution of Higher Professional Education "Smolensk State Medical Academy of Federal Agency of Health Care and Social Development", Smolensk
  - State Institution Scientific Research Institute of Cardiology of Tomsk Research Center of Siberian Branch of Russian Academy of Medical Sciences, Tomsk
  - SibMedCenter LLC, Tomsk
  - Municipal Healthcare Institution "City Clinical Hospital #2", Yaroslavl
  - State Healthcare Institution of Yaroslavl region "Regional Clinical Hosptal", Yaroslavl
  - Municipal Institution "City Clinical Hospital #40", Yekaterinburg
  - State Healthcare Institution "Sverdlovsk Regional Clinical Hospital #1", Yekaterinburg
- Slovakia (3):
  - MEDIKOL s.r.o., Košice
  - SMOLKO s.r.o., Košice
  - FN Trnava, Trnava

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Groups:
- HX575, EPO HEXAL: HX575 recombinant human erythropoietin alfa: Solution for injection (s.c.)
Period: Treatment Period (up to 1 Year)
Arm/Group | HX575, EPO HEXAL | ERYPO
Started | 174 | 163
Completed | 37 | 29
Not Completed | 137 | 134
Period: Safety Follow-up Period (6 Months)
Arm/Group | HX575, EPO HEXAL | ERYPO
Started | 151 (Study terminated prematurely, all available randomized patients followed-up 6 months for safety) | 119 (Study terminated prematurely, all available randomized patients followed-up 6 months for safety)
Completed | 144 | 112
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Treatmen HX575 EPO HEXAL: HX575 recombinant human erythropoietin alfa: Solution for injection (s.c.)
- Treatment ERYPO: ERYPO: Solution for injection (s.c.)
- Total: Total of all reporting groups
Arm/Group | Treatmen HX575 EPO HEXAL | Treatment ERYPO | Total
Number analyzed (Participants) | 174 | 163 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (14.4) | 64.9 (15) | 64.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 98 | 195
  Male | 77 | 65 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 167 | 155 | 322
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Austria | 4 | 1 | 5
  Czech Republic | 22 | 19 | 41
  Russian Federation | 29 | 24 | 53
  Romania | 47 | 52 | 99
  Poland | 13 | 14 | 27
  Slovakia | 4 | 3 | 7
  Bulgaria | 4 | 4 | 8
  France | 0 | 1 | 1
  Germany | 45 | 39 | 84
  India | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin Level
Description: Mean absolute change in hemoglobin (baseline to end of study week 13)
Time Frame: 13 weeks
Population: Full analysis set required: "all randomized patients who received at least one dose of the study medication and for whom at least one Hb value after study day 27 was available". 3 out of 174 patients started in EPO HEXAL group and 6 out of 163 patients started in ERYPO group had no Hb values after study day 27 so they were excluded from analysis.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HX575, EPO HEXAL | ERYPO
Number analyzed (Participants) | 171 | 157
g/dL | 2.2 (1.0) | 2.1 (1.2)

2. Primary Outcome: Weekly Epoetin Dose
Description: Mean weekly epoetin dose [IU/kg] in study weeks 11-13
Time Frame: weeks 11-13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | HX575, EPO HEXAL | ERYPO
Number analyzed (Participants) | 171 | 157
IU/kg | 55.1 (41.9) | 57.9 (46.6)

3. Secondary Outcome: Immunogenicity
Description: Number of participants with antibody formation against Epoetin during treatment period (safety set)
Time Frame: 13 weeks
Measure: Number; unit: participants
Arm/Group | Treatmen HX575 EPO HEXAL | Treatment ERYPO
Number analyzed (Participants) | 174 | 163
participants | 5 | 2

ADVERSE EVENTS:
Time Frame: Treatment period: up to 1 year; Safety follow up period: 6 months
Description: Safety Population (SAF) was composed of all patients who received at least one dose of the study medication during treatment period
Groups:
- Treatment HX575, EPO HEXAL: HX575 recombinant human erythropoietin alfa: Solution for injection (s.c.)
- Safety Follow-up HX575, EPO HEXAL: Patients received HX575, EPO HEXAL during Treatment Period
- Safety Follow-up ERYPO: Patients received ERYPO during Treatment Period
Arm/Group | Treatment HX575, EPO HEXAL | Treatment ERYPO | Safety Follow-up HX575, EPO HEXAL | Safety Follow-up ERYPO
All-Cause Mortality (participants affected / at risk) | 6/174 | 14/163 | 2/151 | 1/119
Serious Adverse Events (participants affected / at risk) | 50/174 | 70/163 | 22/151 | 24/119
Other Adverse Events (participants affected / at risk) | 137/174 | 132/163 | 87/151 | 58/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment HX575, EPO HEXAL (N=174) | Treatment ERYPO (N=163) | Safety Follow-up HX575, EPO HEXAL (N=151) | Safety Follow-up ERYPO (N=119)
Renal failure chronic (Renal and urinary disorders) | 12 (13) | 22 (22) | 11 (11) | 10 (10)
Renal failure (Renal and urinary disorders) | 7 (7) | 6 (6) | 2 (2) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2) | 7 (7) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perianal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertrophy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0
Anti-erythropoietin antibody positive (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mesenteric occlusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment HX575, EPO HEXAL (N=174) | Treatment ERYPO (N=163) | Safety Follow-up HX575, EPO HEXAL (N=151) | Safety Follow-up ERYPO (N=119)
Nasopharyngitis (Infections and infestations) | 17 (23) | 14 (17) | 5 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 16 (21) | 12 (14) | 5 (5) | 6 (7)
Oedema peripheral (General disorders) | 21 (28) | 17 (22) | 4 (4) | 2 (2)
Fatigue (General disorders) | 10 (13) | 1 (1) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 8 (10) | 9 (10) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 38 (73) | 41 (88) | 10 (14) | 10 (11)
Renal failure chronic (Renal and urinary disorders) | 13 (16) | 24 (24) | 13 (13) | 11 (13)
Renal impairment (Renal and urinary disorders) | 3 (3) | 9 (9) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 11 (13) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 4 (4) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 5 (6) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 6 (7) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 7 (7) | 6 (6) | 3 (3) | 2 (2)
Oedema (General disorders) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 6 (6) | 2 (2) | 2 (2)
Asthenia (General disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 6 (7) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 8 (9) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 5 (5) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 5 (6) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (6) | 3 (4) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5) | 5 (6) | 2 (2)
Dizziness (Nervous system disorders) | 7 (7) | 4 (4) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 4 (5) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 1 (1) | 2 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 4 (4) | 4 (4) | 1 (1) | 1 (1)
Anti-erythropoietin antibody positive (Investigations) | 5 (7) | 2 (2) | 5 (5) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 0 (0) | 4 (4) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to the first publication or presentation of the results of the study which is intended to be a joint, multi-center publication of the study results. Following the first publication, institutions and/or Principal Investigators may publish or present data or results from the study per the terms of the clinical trial agreement.